CLINICAL TRIAL: NCT05485363
Title: Non-invasive Assessment of Intracranial Pressure Using Ocular Sonography in Patients Undergoing Laparoscopic Sleeve Gastrectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, MOHAMMED FAWZI ALI ABOSAMAK, Associate professor of anesthesia, intensive care and pain management, Tanta University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1234
Record Dates: First submitted 2022-07-29; First posted 2022-08-03 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: Optic Nerve Sheath Diameter; Laparoscopic Sleeve Gastrectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- optic nerve sheath diameter by using ocular sonography (Experimental)
  Interventions: Diagnostic Test: ultrasonographic measurement of the optic nerve sheath diameter

INTERVENTIONS:
Diagnostic Test: ultrasonographic measurement of the optic nerve sheath diameter — Assessing the optic nerve sheath diameter as an indicator of intracranial pressure during different positions and on specific time intervals in patients undergoing laparoscopic sleeve gastrectomy

SUMMARY:
Laparoscopic gastric sleeve gastrectomy is becoming an increasingly frequent procedure for patients with severe obesity and its related diseases, such as type 2 diabetes, hypertension, dyslipidemia, and sleep apnea.

Assessing the optic nerve sheath diameter (ONSD) with noninvasive ultrasonography has shown to be accurate in determining increased ICP as pressure changes in the subarachnoid space and the cerebrospinal fluid reflect variations in the optic nerve sheath (ONS).

The investigators hypothesized that if ICP during laparoscopy is different according to the position, ONSD would likewise be different. Thus, investigators will investigate the change of ONSD according to the positional change in laparoscopic sleeve gastrectomy surgery.

DETAILED DESCRIPTION:
Laparoscopic gastric sleeve gastrectomy is becoming an increasingly frequent procedure for patients with severe obesity and its related diseases, such as type 2 diabetes, hypertension, dyslipidemia, and sleep apnea.

The impacts of laparoscopy on the intracranial pressure (ICP) are well-documented and several studies have demonstrated that the induction of artificial pneumoperitoneum provokes a measurable increase in ICP. The mechanisms of increase of ICP during laparoscopy are suggested as follows: increase of intra-abdominal pressure, impairment of cerebrospinal fluid (CSF) absorption and impeded drainage of the lumbar venous plexus, increased pressure in the vascular compartment of sacral spaces, Trendelenburg position, and cerebral vasodilation due to hypercarbia.

Neurological comorbidities resulting in chronically elevated ICP-pseudotumor cerebri and idiopathic intracranial hypertension-may develop in morbidly obese individuals without discernable clinical manifestations.

Assessing the optic nerve sheath diameter (ONSD) with noninvasive ultrasonography has shown to be accurate in determining increased ICP as pressure changes in the subarachnoid space and the cerebrospinal fluid reflect variations in the optic nerve sheath (ONS) .

A study on ultrasonographic measurement of ONSD laparoscopic radical prostatectomy with steep Trendelenburg positioning revealed that ONSD increased approximately 12.5% and the increase of ICP corresponding to change of ONSD could be predicted. However, no study measured the changes of ONSD according to the positional change with reversed Trendelenburg position during laparoscopic sleeve gastrectomy. The investigators hypothesized that if ICP during laparoscopy is different according to the position, ONSD would likewise be different. Thus, investigators will investigate the change of ONSD according to the positional change in laparoscopic sleeve gastrectomy surgery.

ELIGIBILITY:
Inclusion Criteria:

* patients older than 18 years old undergoing laparoscopic sleeve gastrectomy under general anesthesia.

Exclusion Criteria:

* pre-existing neurological (e.g. hydrocephalus, intracranial hemorrhage, Etc.) Or cerebrovascular disease, past medical history of ocular pathology or surgery and the use of ketamine and/or succinylcholine during anesthesia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2023-01-01 (Estimated); Study Completion 2023-04-01 (Estimated)

PRIMARY OUTCOMES:
optic nerve sheath diameter | 3 months
  will be measured In the supine position after induction of anesthesia, 3 min after the steep anti-Trendelenburg position (35° incline), 3 min after the steep anti-Trendelenburg position combined with pneumoperitoneum, every 15 minutes and In the supine position after 3 min of de-sufflation of the pneumoperitoneum

SECONDARY OUTCOMES:
Mean blood pressure (MBP) | 3 months
  will be measured In the supine position after induction of anesthesia, 3 min after the steep anti-Trendelenburg position (35° incline), 3 min after the steep anti-Trendelenburg position combined with pneumoperitoneum, every 15 minutes and In the supine position after 3 min of de-sufflation of the pneumoperitoneum
Heart rate (HR) | 3 months
  will be measured In the supine position after induction of anesthesia, 3 min after the steep anti-Trendelenburg position (35° incline), 3 min after the steep anti-Trendelenburg position combined with pneumoperitoneum, every 15 minutes and In the supine position after 3 min of de-sufflation of the pneumoperitoneum
Airway peak pressure (Ppeak) | 3 months
  will be measured In the supine position after induction of anesthesia, 3 min after the steep anti-Trendelenburg position (35° incline), 3 min after the steep anti-Trendelenburg position combined with pneumoperitoneum, every 15 minutes and In the supine position after 3 min of de-sufflation of the pneumoperitoneum
ETCO2 | 3 months
  will be measured In the supine position after induction of anesthesia, 3 min after the steep anti-Trendelenburg position (35° incline), 3 min after the steep anti-Trendelenburg position combined with pneumoperitoneum, every 15 minutes and In the supine position after 3 min of de-sufflation of the pneumoperitoneum

IPD SHARING:
Plan to Share IPD: Undecided